CLINICAL TRIAL: NCT03662165
Title: A Randomised Controlled Trial to Increase HIV Testing Demand Among Truck Drivers and Sex Workers Through Offering Self-Administered Oral HIV Testing at North Star Alliance Clinics in Kenya
Brief Title: Increase HIV Testing Among Truck Drivers and Female Sex Workers in Kenya Through Offering HIV Self-Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City University of New York, School of Public Health (Other)
Collaborators: International Initiative for Impact Evaluation (Other); North Star Alliance (Unknown); University of KwaZulu (Other); New York State Psychiatric Institute (Other)
Responsible Party: Principal Investigator, Elizabeth Kelvin, Associate Professor, City University of New York, School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 2015-0645
Record Dates: First submitted 2018-09-02; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: HIV Testing
Keywords: HIV testing; Truck drivers; sex workers
MeSH Terms: interventions — Methods

STUDY DESIGN:
Intervention Model Description: We selected a sample of eligible truckers and randomized them on a 1:1:1 ratio to the three study arms. After completing the 2 month follow-up, we followed the same procedure with a sample of eligible female sex workers.
Who Masked: Participant
Masking Description: Participants were not informed about the specific research question or the fact that they would be randomized to different HIV testing options in order to avoid bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): The primary intervention consisted of a text message informing participants that HIV self-test kits were available at all North Star Alliance clinics in Kenya. The message was sent three times, one week apart, first in Kiswahili, then in English and then again in Kiswahili, and read: "You can now self-test at home or in the clinic for HIV using a new test kit available from all North Star Alliance clinics in Kenya. Your health, our priority."
  Interventions: Behavioral: Intervention
- Enhanced Standard of Care (Experimental): Those randomized to the enhanced Standard of Care (SOC) arm received the SOC message reminding clients about HIV testing sent three times, one week apart first in Kiswahili, then in English and then again in Kiswahili. The message read: "North Star Alliance East Africa would wish to kindly remind you to visit any of our roadside wellness centres for HIV testing. Your health, our priority."
  Interventions: Behavioral: Enhanced Standard of Care
- Traditional Standard of Care (Active Comparator): Those randomized to the traditional SOC arm received the SOC message one time sent simultaneously in both Kiswahili and English. The message read: "North Star Alliance East Africa would wish to kindly remind you to visit any of our roadside wellness centres for HIV testing. Your health, our priority."
  Interventions: Behavioral: Traditional Standard of Care

INTERVENTIONS:
Behavioral: Intervention — A text was sent three times, one week apart, first in Kiswahili, then in English and then again in Kiswahili, and read: "You can now self-test at home or in the clinic for HIV using a new test kit available from all North Star Alliance clinics in Kenya. Your health, our priority." Participants who came to any North Star clinic in Kenya in the intervention arm were given a demonstration of the self-testing kit and then offered a choice among (1) the standard provider-administered blood-based HIV test; (2) the self-administered oral HIV test for use in the clinic with provider supervision; or (3) the self-administered oral HIV test kit for home use with phone-based post-test counseling.
  Arms: Intervention
Behavioral: Enhanced Standard of Care — Those randomized to the enhanced Standard of Care (SOC) arm received the SOC message reminding clients about HIV testing sent three times, one week apart first in Kiswahili, then in English and then again in Kiswahili. The message read: "North Star Alliance East Africa would wish to kindly remind you to visit any of our roadside wellness centres for HIV testing. Your health, our priority." Participants who came to any North Star clinic in the enhanced SOC arm only offered the standard provider-administered blood-based HIV test.
  Arms: Enhanced Standard of Care
Behavioral: Traditional Standard of Care — Those randomized to the traditional Standard of Care (SOC) arm received the SOC message reminding clients about HIV testing sent one time in both Kiswahili, then in English and Kiswahili simultaneously. The message read: "North Star Alliance East Africa would wish to kindly remind you to visit any of our roadside wellness centres for HIV testing. Your health, our priority." Participants who came to any North Star clinic in the traditional SOC arm only offered the standard provider-administered blood-based HIV test.
  Arms: Traditional Standard of Care

SUMMARY:
The study aimed to assess whether advertising the availability of self-administered oral HIV testing kits increases the number of truck drivers and female sex workers who come to the North Star Alliance clinics for HIV testing (Demand creation). The investigators sent text messages to eligible truck drivers and female sex workers registered in the North Star Alliance electronic health record system who, based on those records, were not accessing HIV testing regularly and randomized them to receive one of two messaged, (1) the standard message sent to all clients who have not tested for HIV in the past 3 months reminding them of the availability of HIV testing at North Star clinics or (2) a text message announcing the availability of HIV self-testing kits fat all North Star clinics in Kenya. The investigators then compared the number of truck drivers and female sex workers from our samples who came to the clinic for HIV testing over a 2 month period following the first text message in the two study arms.

DETAILED DESCRIPTION:
The study aimed to assess whether advertising the availability of self-administered oral HIV testing kits increases the number of truck drivers and female sex workers who come to the North Star Alliance clinics for HIV testing (Demand creation). The investigators first selected a sample of eligible truck drivers from the electronic health record system of the North Star Alliance who, based on those records, were not accessing HIV testing regularly, sent passive text messages alerting them that The North Star Alliance was planning to use their deidentified electronic health data for program evaluation purposes and gave them the option to opt out of being included. The investigators then randomized those who did not opt-out on a 1:1:1 ratio to receive one of two messages, (1) the standard (SOC) message sent to all clients who have not tested for HIV in the past 3 months reminding them of the availability of HIV testing at North Star clinics sent one time (2) the SOC message sent three times, a week apart (Enhanced SOC) or (2) a text message announcing the availability of HIV self-testing kits fat all North Star clinics in Kenya sent three times, a week apart. The investigators compared the number of truck drivers from our sample who came to the clinic for HIV testing over a 2 month period following the first text message in the three study arms. After completing the study among truck drivers, we followed the same procedures for a sample of female sex workers registered in the electronic health record system who were not accessing HIV testing regularly.

ELIGIBILITY:
Inclusion Criteria:

* Truck Drivers or Trucking Assistants (Sample 1) and female sex workers(Sample 2) registered in the North Star Alliance electronic health record system and who
* had no indication that they were HIV-positive
* resided in Kenya
* had a valid mobile phone number listed
* had fewer than four HIV tests recorded in the system in the past 12 months (indicating that they were not following the recommendation to test every 3 months for 4 tests per year), and
* had not had an HIV test in the past 3 months.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4458 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

PRIMARY OUTCOMES:
The Proportion who tested for HIV over 2 months follow-up | 2 months following the first text message
  We compared the proportion who tested for HIV during the 2-month follow-up period among participants in the Intervention arm versus those in the Enhanced Standard of Care (SOC) arm (primary comparison) as well as among those in the Enhanced SOC versus those in the Traditional SOC arms (secondary comparison) to look at the impact of the content of the text message (i.e. about self-testing kits or HIV testing in general) and of the number of text messages (3 versus 1) on HIV testing, respectively.

SECONDARY OUTCOMES:
Proportion who had any clinic contact over the 2 month follow-up | 2 months
  We also looked at differences in clinic contact for any reason (i.e., for HIV testing or some other service) between the three groups to see if the text messages brought more clients to the clinic even if some chose not to test for HIV.
Effect Modification of HIV testing outcome by HIV testing history (Had an HIV test in the past year or not) | 2 months
  We also looked at whether the differences in HIV testing by study arm were modified by HIV testing history (whether the client had an HIV test at a North Star Alliance clinic in the past year).

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Kelvin, PhD, Principal Investigator — City University of New York
Locations (1):
- CUNY Graduate School of Public Health and Health Policy, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All study deidentified data and documentation (e.g. statistical analysis code, study report) has been provided to the study funder (International Initiative for Impact Evaluation) and they will make it publicly available. We will include instructions abut how to access the study data and documents in all publications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: As soon as the main study papers have been accepted fro publication. We have already posted the data from the sex worker sample and will post the data for the trucker sample once the paper has been accepted for publication
Access Criteria: Open access
URL: https://dataverse.harvard.edu/dataset.xhtml?persistentId=doi:10.7910/DVN/UULS6T

REFERENCES:
- [Result] Kelvin EA, George G, Mwai E, Kinyanjui S, Romo ML, Odhiambo JO, Oruko F, Nyaga E, Govender K, Mantell JE. A Randomized Controlled Trial to Increase HIV Testing Demand Among Female Sex Workers in Kenya Through Announcing the Availability of HIV Self-testing Via Text Message. AIDS Behav. 2019 Jan;23(1):116-125. doi: 10.1007/s10461-018-2248-5. PMID 30109456
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Kelvin EA, George G, Kinyanjui S, Mwai E, Romo ML, Oruko F, Odhiambo JO, Nyaga EN, Mantell JE, Govender K. Announcing the availability of oral HIV self-test kits via text message to increase HIV testing among hard-to-reach truckers in Kenya: a randomized controlled trial. BMC Public Health. 2019 Jan 3;19(1):7. doi: 10.1186/s12889-018-6345-1. PMID 30606161
- Available data/document: Individual Participant Data Set — https://dataverse.harvard.edu/dataset.xhtml?persistentId=doi:10.7910/DVN/UULS6T